CLINICAL TRIAL: NCT05460325
Title: A Multi-center, Open-label Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of Lanadelumab (SHP643) in Chinese Subjects With Hereditary Angioedema
Brief Title: A Study of Lanadelumab (SHP643) in Chinese Participants With Hereditary Angioedema (HAE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP643-304
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — lanadelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lanadelumab 300 mg (Experimental): Participants received lanadelumab 300 milligrams (mg), subcutaneously (SC), once every 2 weeks (Q2W) from Day 0 to Day 182 (26 weeks).
  Interventions: Drug: Lanadelumab

INTERVENTIONS:
Drug: Lanadelumab — Lanadelumab subcutaneous injection
  Other Names: SHP643; TAKHZYRO; TAK-743; DX-2930; Lanadelumab Injection

SUMMARY:
The main aim of this study is to evaluate the safety of lanadelumab in Chinese participants with HAE.

Participants will be treated with lanadelumab for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Be of Chinese descent, defined as born in China and having Chinese parents and Chinese maternal and paternal grandparents.
2. The participant is male or female and greater than or equal to (>=) 12 years of age at the time of informed consent.
3. Documented diagnosis of HAE Type I or Type II based upon all of the following:

   * Documented clinical history consistent with HAE (subcutaneous [SC] or mucosal, nonpruritic swelling episodes without accompanying urticaria).
   * Diagnostic testing results obtained during screening by a laboratory (approved by the sponsor) that confirm HAE Type I or Type II: C1 esterase inhibitor (C1-INH) functional level <40% of the normal level. Participants with functional C1-INH level 40% to 50% of the normal level may be enrolled if they also have a C4 level below the normal range. Participants may begin participating in the run-in period before these diagnostic results are available. Participants may be re-tested if results are incongruent with clinical history or believed by the investigator to be confounded by recent long-term prophylaxis (LTP) use.
   * At least one of the following: Age at reported onset of first angioedema symptoms less than or equal to (<=) 30 years, a family history consistent with HAE Type I or Type II, or C1q within normal range.
4. Attack rate:

   • At the time of enrollment, participants must experience at least 1 investigator-confirmed HAE attack per 4 weeks during the run-in period.
5. The participant (or the participant's parent/legal guardian, if applicable) has provided written informed consent approved by the institutional review board (IRB)/ institutional ethical committee (IEC).

   • If the participant is an adult, be informed of the nature of the study and provide written informed consent before any study-specific procedures are performed.

   OR

   • If the participant is a minor (that is <18 years of age), have a parent/legal guardian who is informed of the nature of the study provide written informed consent (that is, permission) for the minor to participate in the study before any study-specific procedures are performed. Assent will be obtained from minor participants.
6. Males, or non-pregnant, non-lactating females who are fertile and sexually active and who agree to be abstinent or agree to comply with the applicable contraceptive requirements of this protocol for the duration of the study, or females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or postmenopausal for at least 12 months.
7. Agree to adhere to the protocol-defined schedule of assessments and procedures.

Exclusion Criteria:

1. Concomitant diagnosis of another form of chronic, recurrent angioedema, such as acquired angioedema, HAE with normal C1 esterase inhibitor (C1-INH) (also known as HAE Type III), idiopathic angioedema, or recurrent angioedema associated with urticaria.
2. Participation in a prior lanadelumab study or use any lanadelumab prior to the study.
3. Dosing with investigational drug or exposure to an investigational device within 4 weeks prior to entering to screening.
4. Exposure to angiotensin-converting enzyme inhibitors or any estrogen-containing medications with systematic absorption (such as oral contraceptives or hormonal replacement therapy) within 4 weeks prior to screening.
5. Exposure to androgens (that is, danazol, methyltestosterone, testosterone) within 2 weeks prior to entering the run-in period.
6. Use of LTP therapy (defined as continued use) for HAE (C1-INH, attenuated androgens, or anti-fibrinolytics) for adult participants within 2 weeks prior to entering the run-in period. Adolescent participants (>=12 to <18 years of age) who are on LTP therapy for HAE are allowed to enter the study.
7. Use of short-term prophylaxis for HAE 7 days prior to entering the run-in period. Short-term prophylaxis is defined as fresh frozen plasma (FFP), C1-INH, attenuated androgens, or antifibrinolytics used to avoid angioedema complications from medically indicated procedures. Note: Currently, C1-INH therapies are not available in China.
8. Any of the following liver function abnormalities: alanine aminotransferase (ALT) greater than (>) 3* upper limit of normal (ULN), or aspartate aminotransferase (AST) > 3* ULN or bilirubin > 2* ULN (unless the bilirubin is a result of Gilbert's syndrome).
9. Pregnancy or breast feeding.
10. Participant has any condition that in the opinion of the investigator or sponsor, may compromise their safety or compliance, preclude successful conduct of the study, or interfere with interpretation of the results (example, history of substance abuse or dependence, significant pre-existing illnesses or major comorbidity the investigator considers may confound the interpretation of the study results).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- China (4):
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Peking Union Medical College Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/43d15f0fe5c54538

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in China from 22 June 2022 to 28 November 2023.
Pre-assignment Details: A total of 20 participants with a diagnosis of hereditary angioedema (HAE) were enrolled in a Run-in Period of 4 to 8 weeks. Participants who experienced ≥1.0 investigator-confirmed HAE attack per 4 weeks during the Run-in Period and who remained eligible per inclusion and exclusion criteria entered the 26-week lanadelumab Treatment Period to receive lanadelumab 300 milligrams (mg).
Groups:
- Lanadelumab 300 mg: Participants received lanadelumab 300 mg, subcutaneously (SC), once every two weeks (Q2W) for 26 weeks.
Period: Run-in Period (4 or up to 8 Weeks)
Arm/Group | Lanadelumab 300 mg
Started | 20
Completed | 20
Not Completed | 0
Period: Treatment Period (Weeks 1 to 26)
Arm/Group | Lanadelumab 300 mg
Started | 20
Completed | 20
Not Completed | 0
Period: Safety Follow-up Period (Weeks 27 to 30)
Arm/Group | Lanadelumab 300 mg
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants who received at least 1 dose of lanadelumab (investigational product [IP]).
Groups:
- Lanadelumab 300 mg: Participants received lanadelumab 300 mg, SC, Q2W for 26 weeks.
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 20
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 67.65 (13.551)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 166.83 (7.973)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)] — BMI = weight (kg)/[height (m)^2]
  kilograms per meter square (kg/m^2) | 24.18 (3.927)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)
Description: TEAE is defined as an adverse event (AE) with onset at the time of or following initial dosing with study drug (lanadelumab), or medical conditions present prior to the start of study drug but increasing in severity or relationship at the time of or following the start of treatment, up to the last follow-up visit. An SAE is any untoward clinical manifestation of signs, symptoms or outcomes whether considered related to investigational product or not and at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, congenital abnormality/birth defect, an important medical event. Hypersensitivity reactions and events of disordered coagulation were considered as AESIs. Adverse events were classified as HAE attack and non-HAE attack reported AEs and are categorized accordingly in this outcome measure. A participant could be counted in more than one category.
Time Frame: From first dose of study drug up to end of study (up to Day 210)
Population: The FAS included all participants who received at least 1 dose of lanadelumab (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
Participants
  TEAEs: Non-Angioedema Attack | 15
  TEAEs: Angioedema Attack | 3
  SAEs: Non-Angioedema Attack | 1
  SAEs: Angioedema Attack | 0
  AESIs: Non-Angioedema Attack | 0
  AESIs: Angioedema Attack | 0

2. Primary Outcome: Number of Participants With Clinically Meaningful Changes in Clinical Laboratory Parameters
Description: Laboratory parameters included clinical chemistry, hematology, coagulation, urinalysis, and serology. Clinically meaningful laboratory parameters assessment was based on investigator interpretation. Number of participants with clinically meaningful changes in laboratory parameters (including clinical chemistry, hematology, coagulation, urinalysis, and serology) were reported.
Time Frame: From first dose of study drug up to end of study (up to Day 210)
Population: The FAS included all participants who received at least 1 dose of lanadelumab (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
Participants | 0

3. Primary Outcome: Number of Participants With Clinically Meaningful Changes in Vital Sign Abnormalities
Description: Vital signs included measurement of blood pressure, heart rate, body temperature, and respiratory rate. Clinically meaningful vital signs assessment was based on investigator interpretation. Number of participants with clinically meaningful changes in vital signs were reported.
Time Frame: From first dose of study drug up to end of study (up to Day 210)
Population: The FAS included all participants who received at least 1 dose of lanadelumab (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
Participants | 0

4. Primary Outcome: Number of Participants With Clinically Meaningful Changes in Electrocardiogram (ECG)
Description: ECG included heart rate, PR interval, QRS duration, QT interval, corrected QT interval (QTc) interval, QT corrected for heart rate by Fridericia's cube root formula (QTcF) interval, and QT corrected for heart rate by Bazett formula (QTcB) interval. Clinically meaningful ECG assessment was based on investigator interpretation. Number of participants with clinically meaningful changes in ECG were reported.
Time Frame: From first dose of study drug up to end of study (up to Day 210)
Population: The FAS included all participants who received at least 1 dose of lanadelumab (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
Participants | 0

5. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Abnormalities on Day 182
Description: Physical examination findings by body system were classified as height and weight, general appearance, ears, nose and throat, head and neck, ophthalmological, respiratory, cardiovascular, abdomen, neurological, extremities, dermatological, and lymphatic. Number of participants with clinically significant changes in physical examination findings per investigator interpretation were reported. Only categories with at least one participant with event are reported.
Time Frame: Day 182
Population: The FAS included all participants who received at least 1 dose of lanadelumab (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
Participants
  Dermatologic System | 2
  Extremities | 1

6. Secondary Outcome: Plasma Concentrations of Lanadelumab
Time Frame: Anytime on Days 0 and 210; and pre-dose on Days 14, 56, 98, 140, 182
Population: The Pharmacokinetic (PK) Set included all participants in the FAS who had at least 1 evaluable post-dose PK concentration value. Number analyzed is the number of participants with data available for analyses at the specified timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
nanograms per milliliter (ng/mL)
  Day 0 | 7.64 (24.096)
  Day 14: Pre-dose: number analyzed (Participants) | 17
  Day 14: Pre-dose | 12336.47 (4531.386)
  Day 56: Pre-dose: number analyzed (Participants) | 19
  Day 56: Pre-dose | 24857.89 (6950.725)
  Day 98: Pre-dose | 24170.00 (7260.426)
  Day 140: Pre-dose: number analyzed (Participants) | 19
  Day 140: Pre-dose | 23821.05 (8808.870)
  Day 182: Pre-dose | 24610.00 (6599.673)
  Day 210 | 12048.00 (3268.807)

7. Secondary Outcome: Plasma Kallikrein (pKal) Activity
Description: pKal activity was measured by cleaved high molecular weight kininogen (cHMWK) level (i.e., plasma concentrations of cHMWK).
Time Frame: Anytime on Days 0 and 210; and pre-dose on Days 14, 56, 98, 140, 182
Population: The Pharmacodynamic (PD) Set included all participants in the FAS who had at least 1 evaluable post-dose PD concentration value. Number analyzed is the number of participants with data available for analyses at the specified timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
ng/mL
  Day 0 | 10256.419 (3311.3810)
  Day 14: Pre-dose: number analyzed (Participants) | 17
  Day 14: Pre-dose | 4904.964 (1350.4121)
  Day 56: Pre-dose: number analyzed (Participants) | 19
  Day 56: Pre-dose | 3604.136 (1279.8551)
  Day 98: Pre-dose | 3312.706 (1526.8282)
  Day 140: Pre-dose: number analyzed (Participants) | 19
  Day 140: Pre-dose | 2871.364 (1324.5022)
  Day 182: Pre-dose | 3383.672 (1337.0341)
  Day 210 | 3800.187 (1499.9735)

8. Secondary Outcome: Number of Investigator-Confirmed HAE Attacks During the Efficacy Evaluation Period of Day 0 Through Day 182
Description: An HAE attack was confirmed by following symptoms or signs consistent with an attack in at least one of the following locations: 1) Peripheral angioedema: cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region; 2) Abdominal angioedema: abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea; 3) Laryngeal angioedema: stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx. Treatment period attack rate per month is calculated as the number of investigator-confirmed HAE attacks occurring during that treatment period divided by number of days the participant contributed to that treatment period multiplied by 28 days.
Time Frame: Day 0 through Day 182
Population: The FAS included all participants who received at least 1 dose of lanadelumab (IP).
Measure: Mean (Standard Deviation); unit: attacks/month
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
attacks/month | 0.04 (0.139)

9. Secondary Outcome: Number of Investigator-Confirmed HAE Attacks That Required Acute Treatment During the Efficacy Evaluation Period of Day 0 Through Day 182
Description: An HAE attack was confirmed by following symptoms/signs consistent with an attack in atleast one of the following locations:1)Peripheral angioedema:cutaneous swelling involving an extremity,the face,neck,torso,and/or genitourinary region;2)Abdominal angioedema:abdominal pain,with/without abdominal distention,nausea,vomiting,or diarrhea;3)Laryngeal angioedema:stridor,dyspnea, difficulty speaking,difficulty swallowing,throat tightening,or swelling of the tongue,palate,uvula,or larynx.Acute HAE attacks were managed per the investigator's usual care, including use of individualized acute therapy/rescue medications.Acute therapy/rescue medications included Firazyr, fresh frozen plasma (FFP), or other local standard of care.Treatment period attack rate per month is calculated as the number of investigator-confirmed HAE attacks requiring acute treatment occurring during that treatment period divided by number of days the participant contributed to that treatment period multiplied by 28 days.
Time Frame: Day 0 through Day 182
Population: The FAS included all participants who received at least 1 dose of lanadelumab (IP).
Measure: Mean (Standard Deviation); unit: attacks/month
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
attacks/month | 0.01 (0.034)

10. Secondary Outcome: Number of Moderate or Severe Investigator-Confirmed HAE Attacks During the Efficacy Evaluation Period of Day 0 Through Day 182
Description: The severity of the investigator-confirmed HAE attacks was defined per the HAE attack assessment and reporting procedures (HAARP) definitions: severe (marked limitation in activity, assistance required), moderate (mild to moderate limitation in activity, some assistance needed). Treatment period attack rate per month is calculated as the number of moderate or severe investigator-confirmed HAE attacks occurring during that treatment period divided by number of days the participant contributed to that treatment period multiplied by 28 days.
Time Frame: Day 0 through Day 182
Population: The FAS included all participants who received at least 1 dose of lanadelumab (IP).
Measure: Mean (Standard Deviation); unit: attacks/month
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
attacks/month | 0.01 (0.034)

11. Secondary Outcome: Number of Participants With Maximum Attack Severity During the Efficacy Evaluation Period of Day 0 Through Day 182
Description: Number of participants with maximum HAE attack severity during the efficacy evaluation period was assessed. HAE attack severity was calculated per participant based on the severity categories as follows: No attack, Mild, Moderate, and Severe.
Time Frame: Day 0 through Day 182
Population: The FAS included all participants who received at least 1 dose of lanadelumab (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
Participants
  No Attack | 18
  Mild | 1
  Moderate | 1
  Severe | 0

12. Secondary Outcome: Time to First Investigator-confirmed HAE Attack During the Efficacy Evaluation Period of Day 0 Through Day 182
Description: Time to the first investigator-confirmed HAE attack (days) was calculated from the date and time of the first dose of study drug for that efficacy evaluation period to the date and time of the first investigator-confirmed HAE attack after the first dose for the efficacy evaluation period. The time to the first HAE attack was summarized using Kaplan-Meier (KM) estimates.
Time Frame: Day 0 through Day 182
Population: The FAS included all participants who received at least 1 dose of lanadelumab (IP).
Measure: Median (Full Range); unit: days
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
days | NA [NA to NA] — Median and full range were not evaluable due to low number of participants with events.

13. Secondary Outcome: Number of Participants Who Achieved Investigator-confirmed HAE Attack-Free Status During the Efficacy Evaluation Period of Day 0 Through Day 182
Description: An HAE attack was confirmed by following symptoms or signs consistent with an attack in at least one of the following locations: 1) Peripheral angioedema: cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region; 2) Abdominal angioedema: abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea; 3) Laryngeal angioedema: stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx. A participant was considered as attack free if the participant had no investigator-confirmed HAE attacks during the efficacy evaluation period. Number of participants who achieved attack-free status for the efficacy evaluation periods were assessed.
Time Frame: Day 0 through Day 182
Population: The FAS included all participants who received at least 1 dose of lanadelumab (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
Participants | 18

14. Secondary Outcome: Number of Participants Who Achieved at Least 50%, 70%, 90%, and 100% Reduction in the Investigator-Confirmed Normalized Number of Attacks (NNA) Per 4 Weeks Relative to the Run-in Period NNA
Description: A run-in period of 4 weeks was included to determine the participant's baseline attack rate. This period may be extended up to 8 weeks. The normalized number of investigator-confirmed HAE attacks during efficacy evaluation period was expressed as a monthly (28 days) HAE attack rate relative to the run-in period NNA. Number of participants who achieved at least 50 percent (%), 70%, 90% and 100% reduction in the investigator-confirmed NNA per 4 weeks relative to the run-in period normalized NNA for the efficacy evaluation periods was assessed.
Time Frame: Day 0 through Day 182
Population: The FAS included all participants who received at least 1 dose of lanadelumab (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
Participants
  ≥50% Reduction | 20
  ≥70% Reduction | 20
  ≥90% Reduction | 19
  100% Reduction | 18

15. Secondary Outcome: Number of Participants Who Achieved NNA <1.0 Per 4 Weeks for the Efficacy Evaluation Period of Day 0 Through Day 182
Description: The normalized number of investigator-confirmed HAE attacks during the efficacy evaluation period was expressed as a monthly (28 days) HAE attack rate. Attack rate was calculated for each participant as the number of attacks occurring during the specified period divided by the number of days the participant contributed to the specified period multiplied by 28 days. Number of participants who achieved NNA <1.0 per 4 weeks for the efficacy evaluation period were assessed.
Time Frame: Day 0 through Day 182
Population: The FAS included all participants who received at least 1 dose of lanadelumab (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
Participants | 20

16. Secondary Outcome: Number of Participants With Neutralizing or Non-neutralizing Antidrug Antibodies (ADA) in Plasma
Description: Number of participants with neutralizing or non-neutralizing ADA in plasma were assessed.
Time Frame: Anytime on Days 0 and 210; and pre-dose on Days 56, 98, 140, 182
Population: The FAS included all participants who received at least 1 dose of lanadelumab (IP). Number analyzed is the number of participants with data available for analyses at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
Participants
  Day 0 | 1
  Day 56: Pre-dose: number analyzed (Participants) | 19
  Day 56: Pre-dose | 0
  Day 98: Pre-dose | 0
  Day 140: Pre-dose: number analyzed (Participants) | 19
  Day 140: Pre-dose | 1
  Day 182: Pre-dose | 1
  Day 210 | 3

17. Secondary Outcome: Plasma Concentrations of Lanadelumab by Immunogenicity Result
Description: The effect of presence or absence of neutralizing or non-neutralizing ADA in plasma on the lanadelumab plasma concentrations was assessed.
Time Frame: Anytime on Days 0 and 210; and pre-dose on Days 56, 98, 140, 182
Population: The PK set included all participants in the FAS who had at least 1 evaluable post-dose PK concentration value. Number analyzed is the number of participants with data available for analyses at the specified timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
ng/mL
  Day 0: Positive ADA Result: number analyzed (Participants) | 1
  Day 0: Positive ADA Result | 0.00 (NA) — Standard deviation (SD) was not estimable for a single participant.
  Day 0: Negative ADA Result: number analyzed (Participants) | 19
  Day 0: Negative ADA Result | 8.04 (24.687)
  Day 56: Pre-dose: Positive ADA Result: number analyzed (Participants) | 0
  Day 56: Pre-dose: Negative ADA Result: number analyzed (Participants) | 19
  Day 56: Pre-dose: Negative ADA Result | 24857.89 (6950.725)
  Day 98: Pre-dose: Positive ADA Result: number analyzed (Participants) | 0
  Day 98: Pre-dose: Negative ADA Result | 24170.00 (7260.426)
  Day 140: Pre-dose: Positive ADA Result: number analyzed (Participants) | 1
  Day 140: Pre-dose: Positive ADA Result | 16700.00 (NA) — SD was not estimable for a single participant.
  Day 140: Pre-dose: Negative ADA Result: number analyzed (Participants) | 18
  Day 140: Pre-dose: Negative ADA Result | 24216.67 (8888.873)
  Day 182: Pre-dose: Positive ADA Result: number analyzed (Participants) | 1
  Day 182: Pre-dose: Positive ADA Result | 27800.00 (NA) — SD was not estimable for a single participant.
  Day 182: Pre-dose: Negative ADA Result: number analyzed (Participants) | 19
  Day 182: Pre-dose: Negative ADA Result | 24442.11 (6736.494)
  Day 210: Positive ADA Result: number analyzed (Participants) | 3
  Day 210: Positive ADA Result | 13800.00 (624.500)
  Day 210: Negative ADA Result: number analyzed (Participants) | 17
  Day 210: Negative ADA Result | 11738.82 (3458.715)

18. Secondary Outcome: Plasma Kallikrein Activity cHMWK by Immunogenicity Result
Description: The effect of presence or absence of neutralizing or non-neutralizing ADA in plasma on the cHMWK levels was assessed.
Time Frame: Anytime on Days 0 and 210; and pre-dose on Days 56, 98, 140, 182
Population: The PD set included all participants in the FAS who had at least 1 evaluable post-dose PD concentration value. Number analyzed is the number of participants with data available for analyses at the specified timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
ng/mL
  Day 0: Positive ADA Result: number analyzed (Participants) | 1
  Day 0: Positive ADA Result | 13346.780 (NA) — SD was not estimable for a single participant.
  Day 0: Negative ADA Result: number analyzed (Participants) | 19
  Day 0: Negative ADA Result | 10093.768 (3319.0248)
  Day 56: Pre-dose: Positive ADA Result: number analyzed (Participants) | 0
  Day 56: Pre-dose: Negative ADA Result: number analyzed (Participants) | 19
  Day 56: Pre-dose: Negative ADA Result | 3604.136 (1279.8551)
  Day 98: Pre-dose: Positive ADA Result: number analyzed (Participants) | 0
  Day 98: Pre-dose: Negative ADA Result | 3312.706 (1526.8282)
  Day 140: Pre-dose: Positive ADA Result: number analyzed (Participants) | 1
  Day 140: Pre-dose: Positive ADA Result | 3733.890 (NA) — SD was not estimable for a single participant.
  Day 140: Pre-dose: Negative ADA Result: number analyzed (Participants) | 18
  Day 140: Pre-dose: Negative ADA Result | 2823.446 (1345.8483)
  Day 182: Pre-dose: Positive ADA Result: number analyzed (Participants) | 1
  Day 182: Pre-dose: Positive ADA Result | 4577.960 (NA) — SD was not estimable for a single participant.
  Day 182: Pre-dose: Negative ADA Result: number analyzed (Participants) | 19
  Day 182: Pre-dose: Negative ADA Result | 3320.814 (1342.9683)
  Day 210: Positive ADA Result: number analyzed (Participants) | 3
  Day 210: Positive ADA Result | 4938.130 (1367.0128)
  Day 210: Negative ADA Result: number analyzed (Participants) | 17
  Day 210: Negative ADA Result | 3599.373 (1467.1561)

19. Secondary Outcome: Number of Investigator-confirmed HAE Attacks by Immunogenicity Result During the Efficacy Evaluation Period of Day 0 Through Day 182
Description: The number of investigator-confirmed HAE attacks during the efficacy evaluation period was expressed as a normalized monthly (4 weeks, i.e., 28 days). Treatment period attack rate per month is calculated as the number of investigator-confirmed HAE attacks occurring during that treatment period divided by number of days the participant contributed to that treatment period multiplied by 28 days. The effect of presence or absence of neutralizing or non-neutralizing ADA in plasma on the investigator-confirmed HAE attacks during the efficacy evaluation period was assessed.
Time Frame: Day 0 through Day 182
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: attacks/month
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 20
attacks/month
  At Least One Positive ADA Result: number analyzed (Participants) | 1
  At Least One Positive ADA Result | 0.00 (NA) — SD was not estimable for a single participant.
  No Positive ADA Result: number analyzed (Participants) | 19
  No Positive ADA Result | 0.04 (0.142)

ADVERSE EVENTS:
Time Frame: From start of the study upto follow up (up to Day 210)
Description: The FAS included all participants who received at least 1 dose of lanadelumab (IP). As per planned analysis, the adverse events were collected in a combined manner (to present under the treatment group of Lanadelumab 300 mg) only for the Treatment Period and Safety follow-up Period.
Arm/Group | Lanadelumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lanadelumab 300 mg (N=20)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lanadelumab 300 mg (N=20)
Abdominal pain upper (Gastrointestinal disorders) | 2
Blood uric acid increased (Investigations) | 2
COVID-19 (Infections and infestations) | 10
Dizziness (Nervous system disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 2
Hypertension (Vascular disorders) | 2
Injection site pain (General disorders) | 4
Injection site swelling (General disorders) | 3
Nasopharyngitis (Infections and infestations) | 2
Nausea (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT05460325/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT05460325/SAP_001.pdf